CLINICAL TRIAL: NCT02250651
Title: The Efficacy and Safety of Bimatoprost SR in Patients With Open-angle Glaucoma or Ocular Hypertension
Brief Title: Efficacy and Safety of Bimatoprost Sustained-Release (SR) in Patients With Open-Angle Glaucoma or Ocular Hypertension
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Allergan (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 192024-092; 2014-003186-24 (EudraCT Number)
Record Dates: First submitted 2014-09-23; First posted 2014-09-26 (Estimated); Results first posted 2021-07-28 (Actual); Last update posted 2021-07-28 (Actual); Status verified 2021-06

CONDITIONS: Glaucoma, Open-Angle; Ocular Hypertension
MeSH Terms: conditions — Glaucoma, Open-Angle; Ocular Hypertension | interventions — Needles; Timolol

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Bimatoprost SR 15 μg (Experimental): Study Eye: bimatoprost sustained-release (SR) 15 micrograms (μg) administered on Day 1 (Period 1), Week 16 (Period 2), and Week 32 (Period 3); timolol vehicle administered once in the morning and once in the evening for up to 20 months. Non-Study Eye: sham administration on Day 1 (Period 1), Week 16 (Period 2), and Week 32 (Period 3); timolol 0.5% administered once in the morning and once in the evening for up to 20 months.
  Interventions: Drug: Bimatoprost SR; Other: Sham: Applicator Without Needle; Drug: Active Comparator: Timolol 0.5%; Drug: Timolol Vehicle (placebo)
- Bimatoprost SR 10 μg (Experimental): Study Eye: bimatoprost SR 10 μg administered on Day 1 (Period 1), Week 16 (Period 2), and Week 32 (Period 3); timolol vehicle administered once in the morning and once in the evening for up to 20 months. Non-Study Eye: sham administration on Day 1 (Period 1), Week 16 (Period 2), and Week 32 (Period 3); timolol 0.5% administered once in the morning and once in the evening for up to 20 months.
  Interventions: Drug: Bimatoprost SR; Other: Sham: Applicator Without Needle; Drug: Active Comparator: Timolol 0.5%; Drug: Timolol Vehicle (placebo)
- Timolol 0.5%: Comparator (Active Comparator): Both Eyes: sham administered on Day 1 (Period 1), Week 16 (Period 2), and Week 32 (Period 3); timolol 0.5% administered once in the morning and once in the evening for up to 20 months.
  Interventions: Other: Sham: Applicator Without Needle; Drug: Active Comparator: Timolol 0.5%

INTERVENTIONS:
Drug: Bimatoprost SR — Bimatoprost SR administered in the study eye on Day 1, Week 16, and Week 32.
  Arms: Bimatoprost SR 10 μg; Bimatoprost SR 15 μg
Other: Sham: Applicator Without Needle — Sham administered on Day 1, Week 16, and Week 32.
Drug: Active Comparator: Timolol 0.5% — Timolol 0.5% administered once in the morning and once in the evening for up to 20 months.
Drug: Timolol Vehicle (placebo) — Timolol vehicle administered once in the morning and once in the evening for up to 20 months.
  Arms: Bimatoprost SR 10 μg; Bimatoprost SR 15 μg

SUMMARY:
This study will evaluate the efficacy and safety of bimatoprost sustained-release (SR) in patients with open-angle glaucoma or ocular hypertension. The study includes a 12-month treatment period with an 8-month extended follow-up.

ELIGIBILITY:
Inclusion Criteria:

- Diagnosis of either open-angle glaucoma or ocular hypertension in each eye and both eyes require IOP-lowering treatment.

Exclusion Criteria:

* Previous enrollment in another Allergan Bimatoprost SR Study
* Eye surgery (including cataract surgery) and/or any eye laser surgery within the past 6 months in the study eye
* Anticipated need for laser eye surgery within the first 52 weeks of the study duration
* History of glaucoma surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 528 (Actual)
Dates: Start 2014-12-15 (Actual); Primary Completion 2018-10-25 (Actual); Study Completion 2020-07-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Margot Goodkin, Study Director — Allergan
Locations (113):
- United States (51):
  - Eye Center South, Dothan, Alabama
  - Arizona Eye Center, Chandler, Arizona
  - Vold Vision, Fayetteville, Arkansas
  - Mark B. Kislinger, MD, Inc., Glendora, California
  - Inland Eye Specialists, Hemet, California
  - Southern California Eye Physicians and Surgeons, Los Alamitos, California
  - Eye Research Foundation, Newport Beach, California
  - North Bay Eye Associates, Inc., Petaluma, California
  - Shasta Eye Medical Group, Inc., Redding, California
  - University of California (UCSF) Department of Ophthalmology, San Francisco, California
  - Pacific Eye Surgeons, San Luis Obispo, California
  - Shepard Eye Center, Santa Maria, California
  - East West Eye Institute, Torrance, California
  - Wolstan & Goldberg Eye Associates, Torrance, California
  - University of Colorado, Aurora, Colorado
  - Insight Vision Group, Parker, Colorado
  - Danbury Eye Physicians and Surgeons PC, Danbury, Connecticut
  - Argus Research at Cape Coral Eye Center, Cape Coral, Florida
  - Specialty Retinal Center, Coral Springs, Florida
  - Bruce A Segal, M.D., Delray Beach, Florida
  - Eye Associates of Fort Myers, Fort Myers, Florida
  - Eye Clinic at Shands Medical Plaza, Gainesville, Florida
  - Bascom Palmer Eye Institute, University of Miami, Palm Beach Gardens, Florida
  - Center for Sight, Sarasota, Florida
  - MedEye Associates, South Miami, Florida
  - Emory University Eye Center, Atlanta, Georgia
  - Virdi Eye Clinic, Rock Island, Illinois
  - Kentuckiana Institute for Eye Research at Bennett & Bloom Eye Centers White House Office Complex, Louisville, Kentucky
  - Johns Hopkins School of Medicine, Wilmer Eye Institute, Baltimore, Maryland
  - Clinical Eye Research of Boston, Co., Winchester, Massachusetts
  - Tekwani Vision Center, St Louis, Missouri
  - Rutgers-New Jersey Medical School, Newark, New Jersey
  - Eye Associates of New Mexico, Albuquerque, New Mexico
  - Mount Sinai School of Medicine, New York, New York
  - Alterman, Modi & Wolter, Poughkeepsie, New York
  - South Shore Eye Care, LLP, Wantagh, New York
  - Charlotte Eye Ear Nose & Throat Associates, PA, Charlotte, North Carolina
  - James D. Branch, MD, Winston-Salem, North Carolina
  - Bergstrom Eye and Laser Clinic, Fargo, North Dakota
  - Legacy Good Samaritan Hospital - Devers Eye Institute, Portland, Oregon
  - Lehigh Valley Eye Center, P.C., Allentown, Pennsylvania
  - Scott & Christie and Associates, PC, Cranberry Township, Pennsylvania
  - Scheie Eye Institute, Department of Ophthalmology, University of Pennsylvania, Philadelphia, Pennsylvania
  - University of Texas Medical Branch, Galveston, Texas
  - Alkek Eye Center, Houston, Texas
  - DCT-Shah Research, LLC dba Discovery ClinicalTrials, Mission, Texas
  - Key Whitman Eye Center, Plano, Texas
  - Vistar Eye Center, Roanoke, Virginia
  - Specialty Eyecare Centre, Bellevue, Washington
  - Wenatchee valley Hospital & Clinics, Clinical research department, Wenatchee, Washington
  - The Eye Centers of Racine and Kenosha, Racine, Wisconsin
- Argentina (8):
  - Instituto Oftalmologico de Buenos Aires Oftalmos, Ciudad Autónoma de Buenos Aires, Buenos Aires
  - Hospital Italiano de Buenos Aires - Hospital, Ciudad Autónoma de Buenos Aires, Buenos Aires
  - Clinica Privada de Ojos, Mar del Plata, Buenos Aires
  - Hospital Universitario Austral, Pilar, Buenos Aires
  - Centro Medico Oftalmologia Global, Rosario, Santa Fe Province
  - Centro Médico Grupo Laser Visión, Rosario, Santa Fe Province
  - Organización Médica de Investigación, Ciudad Autónoma de BuenosAires
  - Oftar Centro Privado de Oftalmologia, Mendoza
- Canada (11):
  - ACS Crichton Prof. Corp, Calgary, Alberta
  - Nova Scotia Health Authority, Department of Ophthalmology & Visual Sciences, Halifax, Nova Scotia
  - Trimed Eye Center, Barrie, Ontario
  - Uptown Eye Specialists, Concord, Ontario
  - Galen Eye Centre, Kingston, Ontario
  - Ophthalmic Consultant Centres Inc, Mississauga, Ontario
  - Sunnybrook Research Institute, Toronto, Ontario
  - Institut De L'Oeil Des Laurentides, Boisbriand, Quebec
  - Clinique d' ophtalmologie Dr Saurel, Drummondville, Quebec
  - Bellevue Clinic, Montreal, Quebec
  - GOGiunta Ophtalmologie, Sherbrooke, Quebec
- Colombia (4):
  - Clinica de Oftalmologia Sandiego S.A., Medellín, Antioquia
  - Fundación Oftalmologica Nacional Fundonal, Bogotá, Bogota D.C.
  - Fundacion Oftalmologica de Santander Foscal, Floridablanca, Santander Department
  - Instituto de Investigaciones, Centro Médico Imbanaco de Cali S.A., Cali
- Czechia (3):
  - Ocni klinika, Brno, Jihlavska
  - Nemocnicni Lekarna, Hradec Králové, Sokolska
  - Ocni klinika Pardubice, Prague
- Egypt (3):
  - Menoufia University Hospital, Shibīn al-Kawm, Cairo Governorate
  - Al Kasr Al Ainy Cairo University Hospital, Cairo
  - Ain Shams University Hospital, Cairo
- Germany (5):
  - Klinikum der Universität Regensburg, Regensburg, Bavaria
  - Augen Zentrum Nordwest, Ahaus, North Rhine-Westphalia
  - Augenärzte am St. Franziskus-Hospital, Münster, North Rhine-Westphalia
  - Universitätsklinik Magdeburg, Magdeburg, Saxony-Anhalt
  - Klinisches Studienzentrum, Mainz
- Italy (6):
  - Università degli Studi G. D'Annunzio Chieti-Pescara, Chieti, Abruzzo
  - Azienda Ospedaliera-Polo Universitario San Paolo, Milan, Lombardy
  - Azienda Ospedaliero Universitaria Policlinico Vittorio Emanuele, Catania, Sicily
  - Oculistica Universitaria Università Degli Studi di Pisa - Ospedale di Cisanello Pisa, Pisa, Tuscany
  - Unità Operativa di Oculistica Ospedale San Raffaele S.r.l., Milan
  - Ospedale Santa Maria Della Misericordia, Perugia
- Hospital Kuala Lumpur Jalan Pahang, Department of Opthalmology, Cheras, Kuala Lumpur, Malaysia
- Capital Eye Specialists, Wellington, New Zealand
- Singapore (3):
  - National University Hospital, Singapore
  - Singapore National Eye Centre, Singapore
  - Changi General Hospital, Singapore
- South Africa (2):
  - Horizon Eye Care Centre, Bloemfontein, Free State
  - Pretoria Eye Institute, Arcadia, Pretoria
- South Korea (3):
  - Seoul National University Hospital, Seoul
  - Samsung Medical Center, Seoul
  - Asan Medical Center, Seoul
- Turkey (Türkiye) (3):
  - Eskisehir Osmangazi Universitesi Goz Hastaliklari Anabilim Dali, Meselik, Eskişehir
  - Marmara Universitesi Pendik Egitim Arastirma Hastanesi Goz Hastaliklari, Pendik, Istanbul
  - Celal Bayar Universitesi Tip Fakultesi Goz Hastaliklari Anabilim Dali, Manisa
- United Kingdom (9):
  - Addenbrookes Hospital, Cambridge
  - Queen Alexandra Hospital, Cosham
  - Princess Alexandra Eye Pavilion, Edinburgh
  - James Paget University Hosp NHS Foundation Trust, Great Yarmouth
  - St Paul's Eye Unit Royal Liverpool&Broadgreen, NHS Trust, Liverpool
  - Aintree University Hospital NHS Foundation Trust, Liverpool
  - ICORG, London
  - In Patient Pharmacy, Ground Floor, Lambeth Wing St Thomas' Hospital, London
  - Peterborough City Hospital Research and Development Department, Peterborough

REFERENCES:
- [Derived] Weinreb RN, Bacharach J, Brubaker JW, Medeiros FA, Bejanian M, Bernstein P, Robinson MR. Bimatoprost Implant Biodegradation in the Phase 3, Randomized, 20-Month ARTEMIS Studies. J Ocul Pharmacol Ther. 2023 Jan-Feb;39(1):55-62. doi: 10.1089/jop.2022.0137. Epub 2022 Nov 15. PMID 36378864
- [Derived] Medeiros FA, Sheybani A, Shah MM, Rivas M, Bai Z, Werts E, Ahmed IIK, Craven ER. Single Administration of Intracameral Bimatoprost Implant 10 microg in Patients with Open-Angle Glaucoma or Ocular Hypertension. Ophthalmol Ther. 2022 Aug;11(4):1517-1537. doi: 10.1007/s40123-022-00527-6. Epub 2022 May 28. PMID 35643967
- [Derived] Bacharach J, Tatham A, Ferguson G, Belalcazar S, Thieme H, Goodkin ML, Chen MY, Guo Q, Liu J, Robinson MR, Bejanian M, Wirta DL; ARTEMIS 2 Study Group. Phase 3, Randomized, 20-Month Study of the Efficacy and Safety of Bimatoprost Implant in Patients with Open-Angle Glaucoma and Ocular Hypertension (ARTEMIS 2). Drugs. 2021 Nov;81(17):2017-2033. doi: 10.1007/s40265-021-01624-9. Epub 2021 Nov 1. PMID 34724172
- See also: More Information — http://www.allerganclinicaltrials.com

RESULTS

PARTICIPANT FLOW:
Groups:
- Timolol 0.5%: Comparator: Study Eye and Non-Study Eye: sham administered on Day 1 (Period 1), Week 16 (Period 2), and Week 32 (Period 3); timolol 0.5% administered once in the morning and once in the evening for up to 20 months.
Period: Treatment Period 1 (Day 1 to Week 15)
Arm/Group | Bimatoprost SR 15 μg | Bimatoprost SR 10 μg | Timolol 0.5%: Comparator
Started | 176 | 176 | 176
Received Sham or Bimatoprost SR | 176 | 175 | 173
Completed | 172 | 170 | 165
Not Completed | 4 | 6 | 11
Not completed — Adverse Event | 0 | 2 | 2
Not completed — Lost to Follow-up | 1 | 0 | 0
Not completed — Personal Reasons | 2 | 3 | 5
Not completed — Protocol Deviation | 1 | 0 | 0
Not completed — Reason not Specified | 0 | 0 | 1
Not completed — Randomized but not Treated | 0 | 1 | 3
Period: Treatment Period 2 (Week 16 to Week 31)
Arm/Group | Bimatoprost SR 15 μg | Bimatoprost SR 10 μg | Timolol 0.5%: Comparator
Started (Started=received administration (Sham or Bimatoprost SR) in the cycle) | 165 | 168 | 165
Completed | 159 | 162 | 160
Not Completed | 6 | 6 | 5
Not completed — Adverse Event | 4 | 1 | 0
Not completed — Lost to Follow-up | 0 | 0 | 3
Not completed — Personal Reasons | 2 | 3 | 2
Not completed — Protocol Deviation | 0 | 1 | 0
Not completed — Reason not Specified | 0 | 1 | 0
Period: Treatment Period 3 (Week 32 to Week 52)
Arm/Group | Bimatoprost SR 15 μg | Bimatoprost SR 10 μg | Timolol 0.5%: Comparator
Started (Started=received administration (Sham or Bimatoprost SR) in the cycle) | 147 | 156 | 159
Completed | 138 | 152 | 154
Not Completed | 9 | 4 | 5
Not completed — Adverse Event | 4 | 1 | 1
Not completed — Lost to Follow-up | 1 | 2 | 1
Not completed — Personal Reasons | 2 | 0 | 2
Not completed — Reason not Specified | 2 | 1 | 1

BASELINE CHARACTERISTICS:
Population: Intent-to-treat (ITT) Population included all randomized participants.
Groups:
- Bimatoprost SR 15 μg: Study Eye: bimatoprost SR 15 μg administered on Day 1 (Period 1), Week 16 (Period 2), and Week 32 (Period 3); timolol vehicle administered once in the morning and once in the evening for up to 20 months. Non-Study Eye: sham administration on Day 1 (Period 1), Week 16 (Period 2), and Week 32 (Period 3); timolol 0.5% administered once in the morning and once in the evening for up to 20 months.
- Total: Total of all reporting groups
Arm/Group | Bimatoprost SR 15 μg | Bimatoprost SR 10 μg | Timolol 0.5%: Comparator | Total
Number analyzed (Participants) | 176 | 176 | 176 | 528
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.8 (10.7) | 62.5 (12.7) | 61.4 (12.4) | 62.6 (12.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 91 | 90 | 88 | 269
  Male | 85 | 86 | 88 | 259
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 116 | 115 | 104 | 335
  Black or African and American | 19 | 20 | 36 | 75
  Asian | 6 | 11 | 13 | 30
  Hispanic | 27 | 22 | 21 | 70
  Other | 8 | 8 | 2 | 18
Intraocular Pressure (IOP) [Mean (Full Range); unit: millimeters of mercury (mmHg)] — IOP is a measurement of the fluid pressure inside the study eye. Measurements were taken at Hours 0 and 2. The study eye is defined as the eye that meets the entry criteria. If both eyes meet the entry criteria, the eye with the higher IOP at Baseline Hour 0 will be selected as the study eye. If both eyes had the same IOP at Hour 0, then the right eye was designated as the study eye. Population: The number analyzed is the number of participants with data available for IOP at Baseline.
  millimeters of mercury (mmHg)
    Hour 0: number analyzed (Participants) | 176 | 176 | 175 | 527
    Hour 0 | 24.39 [18.0 to 32.0] | 24.28 [15.0 to 32.0] | 24.46 [17.0 to 32.0] | 24.38 [15.0 to 32.0]
    Hour 2: number analyzed (Participants) | 176 | 175 | 175 | 526
    Hour 2 | 23.41 [18.5 to 32.0] | 23.24 [14.0 to 32.0] | 23.43 [15.0 to 32.0] | 23.36 [14.0 to 32.0]

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Intraocular Pressure (IOP) in the Study Eye to Week 12 (Hours 0 and 2)
Description: IOP is a measurement of the fluid pressure inside the study eye. Measurements were taken at Hours 0 and 2. The study eye is defined as the eye that meets the entry criteria. If both eyes meet the entry criteria, the eye with the higher IOP at Baseline Hour 0 will be selected as the study eye. If both eyes had the same IOP at Hour 0, then the right eye was designated as the study eye. A mixed-effects model with repeated measures (MMRM) was used for analyses. A negative change from baseline indicates an improvement and a positive change from baseline indicates a worsening.
Time Frame: Baseline (Up to 3 days prior to Day 1 at Hours 0 and 2) to Week 12 (Hours 0 and 2)
Population: Participants from the ITT Population, all randomized participants, with data available for analyses.
Measure: Least Squares Mean (Standard Error); unit: millimeters of mercury (mmHg)
Arm/Group | Bimatoprost SR 15 μg | Bimatoprost SR 10 μg | Timolol 0.5%: Comparator
Number analyzed (Participants) | 176 | 176 | 176
millimeters of mercury (mmHg)
  Change from Baseline at Week 12, Hour 0: number analyzed (Participants) | 168 | 169 | 165
  Change from Baseline at Week 12, Hour 0 | -6.47 (0.30) | -6.18 (0.30) | -6.11 (0.30)
  Change from Baseline at Week 12, Hour 2: number analyzed (Participants) | 168 | 168 | 165
  Change from Baseline at Week 12, Hour 2 | -7.16 (0.28) | -6.72 (0.28) | -6.36 (0.29)
Statistical Analysis 1: Comparison: Bimatoprost SR 15 μg vs Timolol 0.5%: Comparator; Change from Baseline at Week 12, Hour 0: The hypothesis was that bimatoprost SR 15 μg was to be declared non-inferior to timolol 0.5% if the upper limit of the 95% CI was ≤ 1.5 mmHg for all scheduled timepoints (Hours 0 and 2 at Week 12); Test type: Non-Inferiority — MMRM analyses was used with response variable:IOP time-matched change from baseline;Fixed factors: Treatment,timepoint,treatment-by-timepoint interaction and baseline IOP stratification;Covariate:Time-matched baseline IOP and timepoint by time-matched baseline IOP interaction. Unstructured covariance matrix was used; p = 0.3738, MMRM; Least-squares Mean Difference = -0.36, 95% CI 2-sided [-1.17 to 0.44], Standard Error of Mean 0.41
Statistical Analysis 2: Comparison: Bimatoprost SR 10 μg vs Timolol 0.5%: Comparator; Change from Baseline at Week 12, Hour 0: The hypothesis was that bimatoprost SR 10 μg was to be declared non-inferior to timolol 0.5% if the upper limit of the 95% CI was ≤ 1.5 mmHg for all scheduled timepoints (Hours 0 and 2 at Week 12); Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; p = 0.8514, MMRM; Least-squares Mean Difference = -0.08, 95% CI 2-sided [-0.88 to 0.73], Standard Error of Mean 0.41
Statistical Analysis 3: Comparison: Bimatoprost SR 15 μg vs Timolol 0.5%: Comparator; Change from Baseline at Week 12, Hour 2: The hypothesis was that bimatoprost SR 15 μg was to be declared non-inferior to timolol 0.5% if the upper limit of the 95% CI was ≤ 1.5 mmHg for all scheduled timepoints (Hours 0 and 2 at Week 12); Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; p = 0.0401, MMRM; Least-squares Mean Difference = -0.80, 95% CI 2-sided [-1.57 to -0.04], Standard Error of Mean 0.39
Statistical Analysis 4: Comparison: Bimatoprost SR 10 μg vs Timolol 0.5%: Comparator; Change from Baseline at Week 12, Hour 2: The hypothesis was that bimatoprost SR 10 μg was to be declared non-inferior to timolol 0.5% if the upper limit of the 95% CI was ≤ 1.5 mmHg for all scheduled timepoints (Hours 0 and 2 at Week 12); Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; p = 0.3621, MMRM; Least-squares Mean Difference = -0.36, 95% CI 2-sided [-1.12 to 0.41], Standard Error of Mean 0.39

2. Primary Outcome: IOP in the Study Eye at Week 2 (Hour 0)
Description: IOP is a measurement of the fluid pressure inside the study eye. Measurements were taken at Hours 0 and 2. The study eye is defined as the eye that meets the entry criteria. If both eyes meet the entry criteria, the eye with the higher IOP at Baseline Hour 0 will be selected as the study eye. If both eyes had the same IOP at Hour 0, then the right eye was designated as the study eye. MMRM was used for analyses.
Time Frame: Week 2 (Hour 0)
Population: Participants from the ITT Population, all randomized participants, with data available for analyses.
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | Bimatoprost SR 15 μg | Bimatoprost SR 10 μg | Timolol 0.5%: Comparator
Number analyzed (Participants) | 170 | 172 | 172
mmHg | 16.74 (0.27) | 16.92 (0.27) | 17.50 (0.27)
Statistical Analysis 1: Comparison: Bimatoprost SR 15 μg vs Timolol 0.5%: Comparator; Week 2, Hour 0: The hypothesis was that bimatoprost SR 15 μg was to be declared non-inferior to timolol 0.5% if the upper limit of the 95% CI was ≤ 1.5 mmHg for all scheduled timepoints (Hours 0 and 2 at Weeks 2, 6, 12); Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; p = 0.0382, MMRM; Least-squares Mean Difference = -0.76, 95% CI [-1.48 to -0.04], Standard Error of Mean 0.36
Statistical Analysis 2: Comparison: Bimatoprost SR 10 μg vs Timolol 0.5%: Comparator; Week 2, Hour 0: The hypothesis was that bimatoprost SR 10 μg was to be declared non-inferior to timolol 0.5% if the upper limit of the 95% CI was ≤ 1.5 mmHg for all scheduled timepoints (Hours 0 and 2 at Weeks 2, 6, 12); Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; p = 0.1133, MMRM; Least-squares Mean Difference = -0.58, 95% CI [-1.29 to 0.14], Standard Error of Mean 0.36

3. Primary Outcome: IOP in the Study Eye at Week 2 (Hour 2)
Description: as for outcome 2
Time Frame: Week 2 (Hour 2)
Population: Participants from the ITT Population, all randomized participants, with data available for analyses.
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | Bimatoprost SR 15 μg | Bimatoprost SR 10 μg | Timolol 0.5%: Comparator
Number analyzed (Participants) | 170 | 172 | 172
mmHg | 16.09 (0.25) | 16.48 (0.25) | 17.19 (0.25)
Statistical Analysis 1: Comparison: Bimatoprost SR 15 μg vs Timolol 0.5%: Comparator; Week 2, Hour 2: The hypothesis was that bimatoprost SR 15 μg was to be declared non-inferior to timolol 0.5% if the upper limit of the 95% CI was ≤ 1.5 mmHg for all scheduled timepoints (Hours 0 and 2 at Weeks 2, 6, 12); Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; p = 0.0013, MMRM; Least-squares Mean Difference = -1.10, 95% CI [-1.76 to -0.43], Standard Error of Mean 0.34
Statistical Analysis 2: Comparison: Bimatoprost SR 10 μg vs Timolol 0.5%: Comparator; Week 2, Hour 2: The hypothesis was that bimatoprost SR 10 μg was to be declared non-inferior to timolol 0.5% if the upper limit of the 95% CI was ≤ 1.5 mmHg for all scheduled timepoints (Hours 0 and 2 at Weeks 2, 6, 12); Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; p = 0.0364, MMRM; Least-squares Mean Difference = -0.71, 95% CI [-1.38 to -0.05], Standard Error of Mean 0.34

4. Primary Outcome: IOP in the Study Eye at Week 6 (Hour 0)
Description: as for outcome 2
Time Frame: Week 6 (Hour 0)
Population: Participants from the ITT Population, all randomized participants, with data available for analyses.
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | Bimatoprost SR 15 μg | Bimatoprost SR 10 μg | Timolol 0.5%: Comparator
Number analyzed (Participants) | 172 | 171 | 168
mmHg | 17.05 (0.28) | 16.93 (0.28) | 17.51 (0.29)
Statistical Analysis 1: Comparison: Bimatoprost SR 15 μg vs Timolol 0.5%: Comparator; Week 6, Hour 0: The hypothesis was that bimatoprost SR 15 μg was to be declared non-inferior to timolol 0.5% if the upper limit of the 95% CI was ≤ 1.5 mmHg for all scheduled timepoints (Hours 0 and 2 at Weeks 2, 6, 12); Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; p = 0.2304, MMRM; Least-squares Mean Difference = -0.46, 95% CI [-1.22 to 0.29], Standard Error of Mean 0.38
Statistical Analysis 2: Comparison: Bimatoprost SR 10 μg vs Timolol 0.5%: Comparator; Week 6, Hour 0: The hypothesis was that bimatoprost SR 10 μg was to be declared non-inferior to timolol 0.5% if the upper limit of the 95% CI was ≤ 1.5 mmHg for all scheduled timepoints (Hours 0 and 2 at Weeks 2, 6, 12); Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; p = 0.1272, MMRM; Least-squares Mean Difference = -0.59, 95% CI [-1.34 to 0.17], Standard Error of Mean 0.38

5. Primary Outcome: IOP in the Study Eye at Week 6 (Hour 2)
Description: as for outcome 2
Time Frame: Week 6 (Hour 2)
Population: Participants from the ITT Population, all randomized participants, with data available for analyses.
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | Bimatoprost SR 15 μg | Bimatoprost SR 10 μg | Timolol 0.5%: Comparator
Number analyzed (Participants) | 172 | 171 | 168
mmHg | 16.13 (0.26) | 16.53 (0.26) | 17.18 (0.27)
Statistical Analysis 1: Comparison: Bimatoprost SR 15 μg vs Timolol 0.5%: Comparator; Week 6, Hour 2: The hypothesis was that bimatoprost SR 15 μg was to be declared non-inferior to timolol 0.5% if the upper limit of the 95% CI was ≤ 1.5 mmHg for all scheduled timepoints (Hours 0 and 2 at Weeks 2, 6, 12); Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; p = 0.0038, MMRM; Least-squares Mean Difference = -1.05, 95% CI [-1.76 to -0.34], Standard Error of Mean 0.36
Statistical Analysis 2: Comparison: Bimatoprost SR 10 μg vs Timolol 0.5%: Comparator; Week 6, Hour 2: The hypothesis was that bimatoprost SR 10 μg was to be declared non-inferior to timolol 0.5% if the upper limit of the 95% CI was ≤ 1.5 mmHg for all scheduled timepoints (Hours 0 and 2 at Weeks 2, 6, 12); Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; p = 0.0741, MMRM; Least-squares Mean Difference = -0.65, 95% CI [-1.36 to 0.06], Standard Error of Mean 0.36

6. Primary Outcome: IOP in the Study Eye at Week 12 (Hour 0)
Description: as for outcome 2
Time Frame: Week 12 (Hour 0)
Population: Participants from the ITT Population, all randomized participants, with data available for analyses.
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | Bimatoprost SR 15 μg | Bimatoprost SR 10 μg | Timolol 0.5%: Comparator
Number analyzed (Participants) | 168 | 169 | 166
mmHg | 17.39 (0.30) | 17.68 (0.30) | 17.75 (0.30)
Statistical Analysis 1: Comparison: Bimatoprost SR 15 μg vs Timolol 0.5%: Comparator; Week 12, Hour 0: The hypothesis was that bimatoprost SR 15 μg was to be declared non-inferior to timolol 0.5% if the upper limit of the 95% CI was ≤ 1.5 mmHg for all scheduled timepoints (Hours 0 and 2 at Weeks 2, 6, 12); Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; p = 0.3738, MMRM; Least-squares Mean Difference = -0.36, 95% CI [-1.17 to 0.44], Standard Error of Mean 0.41
Statistical Analysis 2: Comparison: Bimatoprost SR 10 μg vs Timolol 0.5%: Comparator; Week 12, Hour 0: The hypothesis was that bimatoprost SR 10 μg was to be declared non-inferior to timolol 0.5% if the upper limit of the 95% CI was ≤ 1.5 mmHg for all scheduled timepoints (Hours 0 and 2 at Weeks 2, 6, 12); Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; p = 0.8514, MMRM; Least-squares Mean Difference = -0.08, 95% CI [-0.88 to 0.73], Standard Error of Mean 0.41

7. Primary Outcome: IOP in the Study Eye at Week 12 (Hour 2)
Description: as for outcome 2
Time Frame: Week 12 (Hour 2)
Population: Participants from the ITT Population, all randomized participants, with data available for analyses.
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | Bimatoprost SR 15 μg | Bimatoprost SR 10 μg | Timolol 0.5%: Comparator
Number analyzed (Participants) | 168 | 169 | 166
mmHg | 16.70 (0.28) | 17.15 (0.28) | 17.50 (0.29)
Statistical Analysis 1: Comparison: Bimatoprost SR 15 μg vs Timolol 0.5%: Comparator; Week 12, Hour 2: The hypothesis was that bimatoprost SR 15 μg was to be declared non-inferior to timolol 0.5% if the upper limit of the 95% CI was ≤ 1.5 mmHg for all scheduled timepoints (Hours 0 and 2 at Weeks 2, 6, 12); Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; p = 0.0401, MMRM; Least-squares Mean Difference = -0.80, 95% CI [-1.57 to -0.04], Standard Error of Mean 0.39
Statistical Analysis 2: Comparison: Bimatoprost SR 10 μg vs Timolol 0.5%: Comparator; Week 12, Hour 2: The hypothesis was that bimatoprost SR 10 μg was to be declared non-inferior to timolol 0.5% if the upper limit of the 95% CI was ≤ 1.5 mmHg for all scheduled timepoints (Hours 0 and 2 at Weeks 2, 6, 12); Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; p = 0.3621, MMRM; Least-squares Mean Difference = -0.36, 95% CI 2-sided [-1.12 to 0.41], Standard Error of Mean 0.39

8. Secondary Outcome: Change From Baseline in IOP in the Study Eye
Description: IOP is a measurement of the fluid pressure inside the study eye. Measurements were taken at Hours 0 and 2. The study eye is defined as the eye that meets the entry criteria. If both eyes meet the entry criteria, the eye with the higher IOP at Baseline Hour 0 will be selected as the study eye. If both eyes had the same IOP at Hour 0, then the right eye was designated as the study eye. MMRM was used for analyses. A negative change from baseline indicates an improvement and a positive change from baseline indicates a worsening.
Time Frame: Baseline (Up to 3 days prior to Day 1 at Hours 0 and 2) to Weeks 2 and 6 (Hours 0 and 2)
Population: Participants from the ITT Population, all randomized participants, with data available for analyses.
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | Bimatoprost SR 15 μg | Bimatoprost SR 10 μg | Timolol 0.5%: Comparator
Number analyzed (Participants) | 176 | 176 | 176
mmHg
  Change from Baseline at Week 2, Hour 0: number analyzed (Participants) | 170 | 172 | 171
  Change from Baseline at Week 2, Hour 0 | -7.12 (0.27) | -6.94 (0.27) | -6.36 (0.27)
  Change from Baseline at Week 2, Hour 2: number analyzed (Participants) | 170 | 171 | 171
  Change from Baseline at Week 2, Hour 2 | -7.77 (0.25) | -7.38 (0.25) | -6.67 (0.25)
  Change from Baseline at Week 6, Hour 0: number analyzed (Participants) | 172 | 171 | 167
  Change from Baseline at Week 6, Hour 0 | -6.81 (0.28) | -6.93 (0.28) | -6.35 (0.29)
  Change from Baseline at Week 6, Hour 2: number analyzed (Participants) | 172 | 170 | 167
  Change from Baseline at Week 6, Hour 2 | -7.74 (0.26) | -7.33 (0.26) | -6.69 (0.27)
Statistical Analysis 1: Comparison: Bimatoprost SR 15 μg vs Timolol 0.5%: Comparator; Change from Baseline at Week 2, Hour 0: The hypothesis was that bimatoprost SR 15 μg was to be declared superior to timolol 0.5% if the upper limit of the 95% CI was <0 mmHg for all scheduled timepoints (Hours 0 and 2 at Weeks 2, 6, 12); Test type: Superiority — [test comment as in outcome 1, analysis 1]; p = 0.0382, MMRM; Least-squares Mean Difference = -0.76, 95% CI 2-sided [-1.48 to -0.04], Standard Error of Mean 0.36
Statistical Analysis 2: Comparison: Bimatoprost SR 10 μg vs Timolol 0.5%: Comparator; Change from Baseline at Week 2, Hour 0: The hypothesis was that bimatoprost SR 10 μg was to be declared superior to timolol 0.5% if the upper limit of the 95% CI was <0 mmHg for all scheduled timepoints (Hours 0 and 2 at Weeks 2, 6, 12); Test type: Superiority — [test comment as in outcome 1, analysis 1]; p = 0.1133, MMRM; Least-squares Mean Difference = -0.58, 95% CI 2-sided [-1.29 to 0.14], Standard Error of Mean 0.36
Statistical Analysis 3: Comparison: Bimatoprost SR 15 μg vs Timolol 0.5%: Comparator; Change from Baseline at Week 2, Hour 2: The hypothesis was that bimatoprost SR 15 μg was to be declared superior to timolol 0.5% if the upper limit of the 95% CI was <0 mmHg for all scheduled timepoints (Hours 0 and 2 at Weeks 2, 6, 12); Test type: Superiority — [test comment as in outcome 1, analysis 1]; p = 0.0013, MMRM; Least-squares Mean Difference = -1.10, 95% CI 2-sided [-1.76 to -0.43], Standard Error of Mean 0.34
Statistical Analysis 4: Comparison: Bimatoprost SR 10 μg vs Timolol 0.5%: Comparator; Change from Baseline at Week 2, Hour 2: The hypothesis was that bimatoprost SR 10 μg was to be declared superior to timolol 0.5% if the upper limit of the 95% CI was <0 mmHg for all scheduled timepoints (Hours 0 and 2 at Weeks 2, 6, 12); Test type: Superiority — [test comment as in outcome 1, analysis 1]; p = 0.0364, MMRM; Least-squares Mean Difference = -0.71, 95% CI 2-sided [-1.38 to -0.05], Standard Error of Mean 0.34
Statistical Analysis 5: Comparison: Bimatoprost SR 15 μg vs Timolol 0.5%: Comparator; Change from Baseline at Week 6, Hour 0: The hypothesis was that bimatoprost SR 15 μg was to be declared superior to timolol 0.5% if the upper limit of the 95% CI was <0 mmHg for all scheduled timepoints (Hours 0 and 2 at Weeks 2, 6, 12); Test type: Superiority — [test comment as in outcome 1, analysis 1]; p = 0.2304, MMRM; Least-squares Mean Difference = -0.46, 95% CI 2-sided [-1.22 to 0.29], Standard Error of Mean 0.38
Statistical Analysis 6: Comparison: Bimatoprost SR 10 μg vs Timolol 0.5%: Comparator; Change from Baseline at Week 6, Hour 0: The hypothesis was that bimatoprost SR 10 μg was to be declared superior to timolol 0.5% if the upper limit of the 95% CI was <0 mmHg for all scheduled timepoints (Hours 0 and 2 at Weeks 2, 6, 12); Test type: Superiority — [test comment as in outcome 1, analysis 1]; p = 0.1272, MMRM; Least-squares Mean Difference = -0.59, 95% CI 2-sided [-1.34 to 0.17], Standard Error of Mean 0.38
Statistical Analysis 7: Comparison: Bimatoprost SR 15 μg vs Timolol 0.5%: Comparator; Change from Baseline at Week 6, Hour 2: The hypothesis was that bimatoprost SR 15 μg was to be declared superior to timolol 0.5% if the upper limit of the 95% CI was <0 mmHg for all scheduled timepoints (Hours 0 and 2 at Weeks 2, 6, 12); Test type: Superiority — [test comment as in outcome 1, analysis 1]; p = 0.0038, MMRM; Least-squares Mean Difference = -1.05, 95% CI 2-sided [-1.76 to -0.34], Standard Error of Mean 0.36
Statistical Analysis 8: Comparison: Bimatoprost SR 10 μg vs Timolol 0.5%: Comparator; Change from Baseline at Week 6, Hour 2: The hypothesis was that bimatoprost SR 10 μg was to be declared superior to timolol 0.5% if the upper limit of the 95% CI was <0 mmHg for all scheduled timepoints (Hours 0 and 2 at Weeks 2, 6, 12); Test type: Superiority — [test comment as in outcome 1, analysis 1]; p = 0.0741, MMRM; Least-squares Mean Difference = -0.65, 95% CI 2-sided [-1.36 to 0.06], Standard Error of Mean 0.36

ADVERSE EVENTS:
Time Frame: First dose of study drug to last visit (Up to approximately 20 months)
Description: All-cause Mortality: Intent-to-treat Population included all randomized participants. Serious and Other Adverse Events (AEs): Safety Population included all participants who received at least 1 administration of study treatment. Ocular AEs reported for Eye Disorders were collected for each eye (study eye or non-study eye [fellow-eye]) separately. The AE footnotes are used to report the number of AEs that occurred in the study eye and in the fellow (non-study) eye.
Arm/Group | Bimatoprost SR 15 μg | Bimatoprost SR 10 μg | Timolol 0.5%: Comparator
All-Cause Mortality (participants affected / at risk) | 1/176 | 0/176 | 1/176
Serious Adverse Events (participants affected / at risk) | 36/176 | 22/175 | 16/173
Other Adverse Events (participants affected / at risk) | 133/176 | 103/175 | 72/173
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | Bimatoprost SR 15 μg (N=176) | Bimatoprost SR 10 μg (N=175) | Timolol 0.5%: Comparator (N=173)
Atrial fibrillation (Cardiac disorders) | 1 | 1 | 0
Myocardial infarction (Cardiac disorders) | 1 | 0 | 1
Angina pectoris (Cardiac disorders) | 1 | 0 | 0
Angina unstable (Cardiac disorders) | 1 | 0 | 0
Coronary artery disease (Cardiac disorders) | 1 | 0 | 0
Supraventricular tachycardia (Cardiac disorders) | 1 | 0 | 0
Cardiac failure congestive (Cardiac disorders) | 0 | 0 | 1
Mitral valve incompetence (Cardiac disorders) | 0 | 0 | 1
Sudden hearing loss (Ear and labyrinth disorders) | 0 | 1 | 0
Ascites (Gastrointestinal disorders) | 1 | 0 | 0
Pancreatitis (Gastrointestinal disorders) | 1 | 0 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 2
Diverticular perforation (Gastrointestinal disorders) | 0 | 0 | 1
Nausea (Gastrointestinal disorders) | 0 | 0 | 1
Death (General disorders) | 0 | 0 | 1
Cholangitis acute (Hepatobiliary disorders) | 1 | 0 | 0
Cholelithiasis (Hepatobiliary disorders) | 0 | 1 | 0
Sarcoidosis (Immune system disorders) | 1 | 0 | 0
Pneumonia (Infections and infestations) | 3 | 0 | 0
Appendicitis (Infections and infestations) | 1 | 0 | 0
Jaw fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Procedural pain (Injury, poisoning and procedural complications) | 1 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 2 | 0
Hip fracture (Injury, poisoning and procedural complications) | 0 | 1 | 1
Femur fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Humerus fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Rib fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Subdural haematoma (Injury, poisoning and procedural complications) | 0 | 1 | 0
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 1 | 0 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Metabolic acidosis (Metabolism and nutrition disorders) | 0 | 0 | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 3 | 0 | 0
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Haemarthrosis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2/85 | 0/85 | 1/88 — Number of participants at risk are male participants as this adverse event is specific to males.
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0 | 0
Breast cancer stage I (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Hepatocellular carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Metastases to liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Metastases to lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Natural killer-cell leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Waldenstrom's macroglobulinaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Bronchial carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Oropharyngeal squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Follicular thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Small intestine carcinoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Encephalopathy (Nervous system disorders) | 1 | 0 | 0
Transient ischaemic attack (Nervous system disorders) | 0 | 2 | 0
Ischaemic stroke (Nervous system disorders) | 0 | 1 | 0
Bipolar disorder (Psychiatric disorders) | 0 | 1 | 0
Depression (Psychiatric disorders) | 0 | 0 | 1
Schizophrenia (Psychiatric disorders) | 0 | 0 | 1
End stage renal disease (Renal and urinary disorders) | 0 | 1 | 0
Acute kidney injury (Renal and urinary disorders) | 0 | 0 | 1
Micturition urgency (Renal and urinary disorders) | 0 | 0 | 1
Nephrolithiasis (Renal and urinary disorders) | 0 | 0 | 1
Menorrhagia (Reproductive system and breast disorders) | 0/91 | 1/90 | 0/85 — Number of participants at risk are female participants as this adverse event is specific to females.
Ovarian cyst (Reproductive system and breast disorders) | 0/91 | 1/90 | 0/85 — Number of participants at risk are female participants as this adverse event is specific to females.
Aortic stenosis (Vascular disorders) | 0 | 1 | 0
Penetrating aortic ulcer (Vascular disorders) | 0 | 0 | 1
Peripheral arterial occlusive disease (Vascular disorders) | 0 | 0 | 1
Corneal endothelial cell loss (Eye disorders) | 9 | 3 | 0 — 12 adverse events occurred in the study eye: (Bimatoprost SR 15 ug=9, Bimatoprost SR 10 ug=3).
Corneal oedema (Eye disorders) | 2 | 1 | 0 — 3 adverse events occurred in the study eye: (Bimatoprost SR 15 ug=2, Bimatoprost SR 10 ug=1).
Macular oedema (Eye disorders) | 1 | 0 | 0 — 1 adverse event occurred in the study eye.
Product administered at inappropriate site (Injury, poisoning and procedural complications) | 1 | 0 | 0
Pterygium (Eye disorders) | 1 | 0 | 0 — 1 adverse event occurred in the study eye.
VIth nerve paralysis (Nervous system disorders) | 1 | 0 | 0
Corneal decompensation (Eye disorders) | 0 | 1 | 0 — 1 adverse event occurred in the study eye.
Retinal detachment (Eye disorders) | 0 | 1 | 0 — 1 adverse event occurred in the study eye.
Visual impairment (Eye disorders) | 0 | 1 | 0 — 1 adverse event occurred in the study eye.
Retinal tear (Eye disorders) | 1 | 0 | 0 — 1 adverse event occurred in the fellow (non-study) eye.
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Bimatoprost SR 15 μg (N=176) | Bimatoprost SR 10 μg (N=175) | Timolol 0.5%: Comparator (N=173)
Conjunctival hyperaemia (Eye disorders) | 73 | 48 | 20 — 138 adverse events occurred in the study eye: (Bimatoprost SR 15 ug=71, Bimatoprost SR 10 ug=48, and Timolol 0.5%=19); 86 adverse events occurred in the fellow (non-study) eye.
Corneal endothelial cell loss (Eye disorders) | 38 | 12 | 2 — 50 adverse events occurred in the study eye: (Bimatoprost SR 15 ug=38, Bimatoprost SR 10 ug=11, and Timolol 0.5%=1); 4 adverse events occurred in the fellow (non-study) eye.
Eye pain (Eye disorders) | 23 | 12 | 9 — 40 adverse events occurred in the study eye: (Bimatoprost SR 15 ug=21, Bimatoprost SR 10 ug=11, and Timolol 0.5%=8); 16 adverse events occurred in the fellow (non-study) eye.
Corneal oedema (Eye disorders) | 21 | 5 | 0 — 26 adverse events occurred in the study eye: (Bimatoprost SR 15 ug=21, Bimatoprost SR 10 ug=5).
Foreign body sensation in eyes (Eye disorders) | 19 | 18 | 2 — 37 adverse events occurred in the study eye: (Bimatoprost SR 15 ug=18, Bimatoprost SR 10 ug=17, and Timolol 0.5%=2); 17 adverse events occurred in the fellow (non-study) eye.
Dry eye (Eye disorders) | 18 | 12 | 7 — 33 adverse events occurred in the study eye: (Bimatoprost SR 15 ug=16, Bimatoprost SR 10 ug=10, and Timolol 0.5%=7); 31 adverse events occurred in the fellow (non-study) eye.
Conjunctival haemorrhage (Eye disorders) | 17 | 20 | 15 — 42 adverse events occurred in the study eye: (Bimatoprost SR 15 ug=14, Bimatoprost SR 10 ug=16, and Timolol 0.5%=12); 22 adverse events occurred in the fellow (non-study) eye.
Punctate keratitis (Eye disorders) | 14 | 10 | 8 — 28 adverse events occurred in the study eye: (Bimatoprost SR 15 ug=13, Bimatoprost SR 10 ug=8, and Timolol 0.5%=7); 26 adverse events occurred in the fellow (non-study) eye.
Photophobia (Eye disorders) | 13 | 13 | 0 — 26 adverse events occurred in the study eye: (Bimatoprost SR 15 ug=13, Bimatoprost SR 10 ug=13); 13 adverse events occurred in the fellow (non-study) eye.
Eye irritation (Eye disorders) | 13 | 10 | 9 — 28 adverse events occurred in the study eye: (Bimatoprost SR 15 ug=12, Bimatoprost SR 10 ug=9, and Timolol 0.5%=7); 23 adverse events occurred in the fellow (non-study) eye.
Anterior chamber cell (Eye disorders) | 13 | 6 | 1 — 19 adverse events occurred in the study eye: (Bimatoprost SR 15 ug=12, Bimatoprost SR 10 ug=6, and Timolol 0.5%=1); 1 adverse event occurred in the fellow (non-study) eye.
Ocular discomfort (Eye disorders) | 11 | 3 | 1 — 15 adverse events occurred in the study eye: (Bimatoprost SR 15 ug=11, Bimatoprost SR 10 ug=3, and Timolol 0.5%=1); 4 adverse events occurred in the fellow (non-study) eye.
Iritis (Eye disorders) | 9 | 8 | 0 — 17 adverse events occurred in the study eye: (Bimatoprost SR 15 ug=9, Bimatoprost SR 10 ug=8); 1 adverse event occurred in the fellow (non-study) eye.
Lacrimation increased (Eye disorders) | 9 | 7 | 1 — 16 adverse events occurred in the study eye: (Bimatoprost SR 15 ug=9, Bimatoprost SR 10 ug=6, and Timolol 0.5%=1); 12 adverse events occurred in the fellow (non-study) eye.
Vision blurred (Eye disorders) | 7 | 11 | 1 — 17 adverse events occurred in the study eye: (Bimatoprost SR 15 ug=7, Bimatoprost SR 10 ug=9, and Timolol 0.5%=1); 11 adverse events occurred in the fellow (non-study) eye.
Blepharitis (Eye disorders) | 7 | 10 | 5 — 21 adverse events occurred in the study eye: (Bimatoprost SR 15 ug=7, Bimatoprost SR 10 ug=9, and Timolol 0.5%=5); 18 adverse events occurred in the fellow (non-study) eye.
Nasopharyngitis (Infections and infestations) | 9 | 12 | 14
Intraocular pressure increased (Investigations) | 17 | 15 | 6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
A disclosure restriction on the PI is that the sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period that is less than or equal to 90 days from the time submitted to the sponsor for review. The sponsor cannot require changes to the communication and cannot extend the embargo.

DOCUMENTS (2):
  • Study Protocol (2018-06-05): https://cdn.clinicaltrials.gov/large-docs/51/NCT02250651/Prot_000.pdf
  • Statistical Analysis Plan (2018-10-29): https://cdn.clinicaltrials.gov/large-docs/51/NCT02250651/SAP_001.pdf